CLINICAL TRIAL: NCT06024824
Title: DP-IMRT Pancreas: A Non-randomised Phase I/II Study of Dose-escalated Hypofractionated Dose-Painted Intensity Modulated Radiotherapy (DPIMRT) in Resectable/Borderline Resectable Pancreatic Adenocarcinoma
Brief Title: Dose-Painted Intensity Modulated Radiotherapy Pancreas (DP-IMRT Pancreas)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 17-12
Record Dates: First submitted 2023-06-16; First posted 2023-09-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Adenocarcinoma

STUDY DESIGN:
Masking Description: This is a prospective non-randomised Phase I/II Radiotherapy (RT) study with patients recruited to escalated dose cohorts. Patients with resectable or borderline resectable (per the National Comprehensive Cancer Network (NCCN) criteria) pancreatic adenocarcinoma will receive dose-escalated hypofractionated DP-IMRT via Intensity Modulated Radiotherapy (IMRT) / Volume Modulated Arc Therapy (VMAT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation; IMRT (Experimental): Fifteen fractions of external beam radiation therapy (EBRT) delivered via IMRT/ VMAT. Cohort 1 (n = 3-6) Single PTV 40.05 Gy/15#, homogenous dose* Cohort 2 (n = 3-6) High Risk PTV 45 Gy/15# SIB to PTV tumour, Elective PTV 40.05 Gy/15# to nodal regions* Cohort 3 (n = 3-6) High risk PTV 48 Gy/15# SIB to PTV tumour, Elective PTV 40.05 Gy/15# to nodal regions
  * Progression to the next dose in successive cohorts depends on the number of patients experiencing DLTs within 4 weeks post-RT treatment in each patient cohort.
  Interventions: Radiation: Dose-Painted Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Dose-Painted Intensity Modulated Radiotherapy — Fifteen fractions of external beam radiation therapy (EBRT) delivered via IMRT/ VMAT.
  Cohort 1 (n = 3-6) Single PTV 40.05 Gy/15#, homogenous dose. Cohort 2 (n = 3-6) High Risk PTV 45 Gy/15# SIB to PTV tumour, Elective PTV 40.05 Gy/15# to nodal regions.
  Cohort 3 (n = 3-6) High risk PTV 48 Gy/15# SIB to PTV tumour, Elective PTV 40.05 Gy/15# to nodal regions.

SUMMARY:
This is a prospective non-randomised Phase I/II Radiotherapy (RT) study with patients recruited to escalated dose cohorts. Patients with resectable or borderline resectable (per the National Comprehensive Cancer Network (NCCN) criteria) pancreatic adenocarcinoma will receive dose-escalated hypofractionated DP-IMRT via Intensity Modulated Radiotherapy (IMRT) / Volume Modulated Arc Therapy (VMAT).

DETAILED DESCRIPTION:
The study treatment is radiotherapy. Different doses of radiotherapy will be given to patients. The first group of patients will receive the lowest dose (dose level 1) (this is the dose delivered to patients as standard of care). If the treatment does not cause serious side effects, it will be given to the next group of patients enrolled at a higher dose (dose level 2) (this is called 'dose escalation'). If this higher dose of treatment does not cause serious side effects, the next group of patients will receive a higher dose (dose level 3). The doses will continue to increase for every group of patients, as long as no serious side effects occur. If this happens, the study is halted. Once the optimum dose level has been reached, a larger cohort of patients will all receive this dose.

Phase I: A 3+3 dose escalation design is proposed to determine the maximum tolerated dose (MTD) defined by the number of radiotherapy-related ≥ Grade 3 acute toxicities assessed up to 4 weeks post RT. Three cohorts of between 3 and 6 patients at each dose level will be accrued in order to establish the MTD (minimum of 6, maximum of 18 patients). The MTD defined in Phase I will be the dose which will be used in Phase II of the trial. Phase II: 49 patients: Once the MTD is established, patients will continue to be recruited at that dose level up to a total of 49 patients.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent obtained prior to any study-related procedures
2. Age ≥18 years
3. ECOG (European Cooperative Oncology Group) performance status (PS) 0-2
4. Resectable or borderline resectable per National Comprehensive Cancer Network (NCCN) criteria (see Appendix H)
5. Patients with histologically confirmed Pancreatic Ductal Adenocarcinoma (PDAC), with the following staging: cT1N0-2, cT2N0-2, cT3N0-2 [American Joint Committee on Cancer (AJCC) 8th edition] (see Appendix C) who are planned for pre-operative systemic chemo-radiotherapy
6. Imaging with Computed Tomography Thorax Abdomen and Pelvis (CT TAP) and Magnetic resonance imaging (MRI) Abdomen confirms no evidence of metastatic disease
7. Females of child-bearing potential (see Appendix G) must not be pregnant (or lactating) and must be prepared to use adequate contraception methods during treatment. Males whose female partners are of child-bearing potential must be prepared to use adequate contraception methods during treatment.

Exclusion Criteria

1. Previous thoracic or abdominal or pelvic radiation therapy (RT)
2. Previous treatment for bilirubin regression, other than stenting
3. Known co-existing or prior malignancy within the last 5 years (except for Basal Cell Carcinoma (BCC) or Squamous Cell Carcinoma (SCC) of the skin) which is likely to interfere with treatment or assessment of outcomes
4. Syndromes or conditions associated with increased radiosensitivity
5. Uncontrolled intercurrent illness that is likely to interfere with treatment or assessment of outcomes, or psychiatric illness/ social situations that would limit compliance with study requirements
6. Evidence of any other significant clinical disorder or laboratory findings that makes it undesirable for the patient to participate in the study, or if it is felt by the research/ Medical team that the patient may not be able to comply with the protocol and follow up schedule due to psychological, familial, sociological or geographical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Phase 1 - to establish the MTD in a dose-escalated and hypofractionated RT regime delivered via IMRT/VMAT by the number of DLTs | 4 weeks
  To establish the MTD in a dose-escalated and hypofractionated RT regime delivered via IMRT/VMAT by the number of DLTs, and the rate of patient withdrawal from trial treatment due to DLTs. Analysis will be performed for each cohort after all patients have been assessed for their 4-week post RT assessment.
Phase 2 - to determine the frequency and severity of DLTs due to AE/Toxicity meeting definition of DLT at 4 weeks post RT | 4 weeks
  The rate of DLTs up to 4 weeks post RT will be calculated. This proportion along with the 90% confidence intervals will be reported.
Phase 2 - to determine the rate of patient withdrawal from trial treatment due to AE/Toxicity meeting definition of DLT at 4 weeks post RT | 4 weeks
  The rate of withdrawal from trial treatment of patients due to DLTs will be calculated. This proportion along with the 90% Confidence Interval will be reported. Other toxicity data including SAEs will be summarised and presented in tabular format with proportions plus 95% Confidence Interval where appropriate.

SECONDARY OUTCOMES:
To quantify the percentage of histologically proven R0 resections in the trial patient group (R0 to be defined as a minimal clearance of at least1 mm). | 2 years
  The percentage of histologically proven R0 resections in this patient group (R0 to be defined as a minimal clearance of at least 1 mm) will be presented with 95% Confidence Interval.
To determine the rate of failure to progress to surgery due to disease progression during neoadjuvant radiotherapy, and conversely the proportion of patients who do receive surgical resection | 2 years
  The rate of failure to progress to surgery due to disease progression during neoadjuvant radiotherapy will be presented with 95% Confidence Interval. The rate of progression to surgery will be presented with 95% CI. The proportion of patients who receive surgical resection overall will be presented with 95% Confidence Interval.
To document the proportion of peri-operative complications | 2 years
  The proportion of patients with peri-operative complications will be presented with 95% Confidence Interval.
To evaluate the impact of treatment on OS, overall and by resectability (whether resectable or borderline resectable) | 2 years
  The Kaplan-Meier method will be used to estimate OS. This will be expressed as median survival with 95% Confidence Interval and will be analysed after patients have been followed for two years after completion of study treatment. The Log-rank test will be used to compare differences in survival between resectable and borderline resectable patients.
To evaluate the impact of treatment on PFS, overall and by resectability (whether resectable or borderline resectable) | 2 years
  The Kaplan-Meier method will be used to estimate PFS. This will be expressed as median survival with 95% Confidence Interval and will be analysed after patients have been followed for two years after completion of study treatment. The Log-rank test will be used to compare differences in survival between resectable and borderline resectable patients.
To evaluate tumour response on surgically resected patients using resected specimens | 2 years
  The proportion of surgically resected patients receiving at least 14 fractions of RT with tumour response using the resected specimens will be presented with 95% Confidence Interval.
To evaluate Quality of Life | 2 years
  The mean (and standard deviation) of the overall and domain specific European Organisation for Research and Treatment for Cancer (EORTC) Quality Life Questionnaire (QLQ) C30 scores at each time point will be reported (pre-chemotherapy, pre-RT, pre-surgery, 6-, 12- and 24-months post RT).
  The EORTC QLQ C30 questionnaire has five functioning subscale scores and nine symptoms subscale scores.
  Minimum value = 0; Max value = 100 Function Scales: Higher numbers mean better function Symptom Scale: Higher numbers mean more symptoms
To evaluate Quality of Life | 2 years
  The mean (and standard deviation) of the overall and domain specific European Organisation for Research and Treatment for Cancer (EORTC) Quality Life Questionnaire (QLQ) PAN 26 scores at each time point will be reported (pre-chemotherapy, pre-RT, pre-surgery, 6-, 12- and 24-months post RT).
  The EOTRC QLQ PAN 26 questionnaire is a tumour specific quality of life questionnaire for patients with pancreatic cancer.
  Minimum value = 0; Max value = 100 Function Scales: Higher numbers mean better function Symptom Scale: Higher numbers mean more symptoms
To evaluate the incidence of late GI toxicities in patients who do not undergo surgical resection | 2 years
  The incidence of late toxicity at 6-, 12- and 24-months post-RT, in patients who do not undergo surgical resection, will be calculated, summarised and presented in tabular format with proportions plus 95% Confidence Interval where appropriate. Toxicities of ≥ Grade 2 are of specific interest. Counts and frequencies will be provided for the worst grade AE experienced

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - St Luke's Radiation Oncology Network (SLRON), Dublin
  - St Vincent's University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No